CLINICAL TRIAL: NCT06007612
Title: Context Sensitivity in Emotion Regulation in Post-Traumatic Stress Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gal Sheppes (Other)
Responsible Party: Sponsor-Investigator, Gal Sheppes, Principal Investigator of Emotion Regulation Lab, Tel Aviv University
Organization: Tel Aviv University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Sheppes02
Record Dates: First submitted 2023-08-17; First posted 2023-08-23 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2023-08

CONDITIONS: Complex Post-Traumatic Stress Disorder
Keywords: EMOTION REGULATION
MeSH Terms: conditions — Emotional Regulation

STUDY DESIGN:
Intervention Model Description: 2 groups enrolled in a one-time behavioral paradigm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Behavioral: Context Sensitivity in Emotion Regulation (Experimental)
  Interventions: Behavioral: Context Sensitivity in Emotion Regulation

INTERVENTIONS:
Behavioral: Context Sensitivity in Emotion Regulation — Context Sensitivity of affective intensities and its association to Emotion Regulation Flexibility Selection

SUMMARY:
This study will examine context sensitivity, composed of two sequential elements: (a) accurate classification of changing affective contextual demands, followed by (b) flexible selection of regulatory strategies that matches changing contextual demands, among complex PTSD vs. Healthy controls.

DETAILED DESCRIPTION:
The study will recruit adults with posttraumatic stress disorder (PTSD) due to a repetitive inter-personal trauma and healthy adult controls which do not meet DSM-5 criteria for PTSD and do not meet the clinical cutoff of Anxiety and Depression screening questionnaires.

A compatibility check, filtering, verification of exclusion criteria and informed consent will occur via online self-report questionnaires.

Clinical questioners include:

Life event Checklist (LEC) - PTSD criteria A Post-trauma Checklist for DSM-5 (PCL) - PTSD symptoms Patient Health Questionnaire (PHQ-9) - Depression Symptoms General Anxiety Disorder Questioner (GAD-7) - Anxiety Symptoms

Participants who pass the initial filtering, will be called and provided with an explanation about the study following which they received the online experiment.

Modified regulatory selection flexibility paradigm- included 3 blocks:

(A) Stimuli Classification- 80 emotional words (equally distributed between high or low intensities) are presented and participants are asked classify each emotional word to high or low intensity.

(B) Regulatory Selection- 40 emotional words (out of the 80 presented in block A) are presented and participants are instructed to behaviorally choose between distraction and reappraisal.

(B) Regulatory Selection- 40 emotional words (the 40 remaining from block A) are presented, prior to regulatory selection, participants received accurate normed intensity classification of the word and then participants are instructed to behaviorally choose between distraction and reappraisal.

ELIGIBILITY:
Inclusion Criteria:

* Native Hebrew speakers
* age between 18 - 65
* normal or corrected to normal vision
* computer and internet access
* Group 1: Diagnosis of PTSD according to the DSM-5
* Group 2: GAD and PHQ scores (score<10), no diagnosis of PTSD according to the DSM-5

Exclusion Criteria:

* Psychosis
* substance dependence or abuse other than nicotine
* Neurological condition

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2023-04-13 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Difference in accurate intensity classification measured during Block A of the experiment | During the experimental task (1 hour)
  comparing the accuracy in intensity classification of 80 words stimuli between the PTSD group and the control group.
regulatory selection flexibility (distraction choice in high intensity minus distraction choice in low intensity) as assessed by regulatory selection paradigm | During the experimental task (1 hour)
  group comparison of the association between accuracy in intensity classification (as measured in Block A) and regulatory selection flexibility (measured by the flexibility score which is calculated by subtracting the proportion of distraction selection in the low intensity stimuli (which reflects maladaptive behavior) from the proportion of distraction selection in the high intensity pictures (which reflects adaptive behavior) measured in Block B.
regulatory selection flexibility (measured by distraction choice in high intensity minus distraction choice in low intensity) following provided intensity as assessed by regulatory selection paradigm | During the experimental task (1 hour)
  group comparison of the association between provided intensity classification (i.e., whether stimuli is of high or low intensity) and regulatory selection flexibility (measured by the flexibility score which is calculated by subtracting the proportion of distraction selection in the low intensity stimuli (which reflects maladaptive behavior) from the proportion of distraction selection in the high intensity pictures (which reflects adaptive behavior) measured in Block C

CONTACTS AND LOCATIONS:
Locations (1):
- Tel Aviv University, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: Undecided